CLINICAL TRIAL: NCT02888431
Title: Correlation of Arterial and Venous Lactate and Base Deficit Values
Status: Completed | Type: Observational
Sponsor: Joseph D. Tobias (Other)
Responsible Party: Sponsor-Investigator, Joseph D. Tobias, Chairman, Professor of Anesthesiology, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Other Study IDs: IRB15-00793
Record Dates: First submitted 2016-08-17; First posted 2016-09-05 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Arterial Access; Peripheral Access; Central Venous Catheter
Keywords: pH; base deficit; lactate values; venous blood samples; arterial blood samples

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Arterial blood sample: 0.5 mL blood sample from arterial line which is clinically indicated
  Interventions: Device: bedside point-of-care device
- peripheral venous blood sample: 0.5 mL blood sample drawn simultaneously with arterial sample from clinically indicated peripheral line
  Interventions: Device: bedside point-of-care device

INTERVENTIONS:
Device: bedside point-of-care device — A bedside point-of-care device is routinely used in the operating room to measure lactate, base deficit, and pH.

SUMMARY:
The purpose of this study is to determine the correlation between pH, base deficit, and lactate values when comparing venous and arterial blood samples in the pediatric population.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring arterial access and peripheral access. Additionally, patients with a central venous catheter would be included.

Exclusion Criteria:

* Patients who not require arterial access.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients requiring arterial access and peripheral access. Additionally, patients with a central venous catheter would be included.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2015-09; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
lactate blood value | During surgery- approximately 15-20 minutes after induction in the operating room (OR)
  blood will be drawn from peripheral venous line, arterial line, and/or central venous line then the lactate value will be assessed by using a bedside point-of-care device, called i-stat.
base deficit blood value | During surgery- approximately 15-20 minutes after induction in the operating room (OR)
  blood will be drawn from peripheral venous line, arterial line, and/or central venous line then the base deficit blood value will be assessed by using a bedside point-of-care device, called i-stat.
pH blood value | During surgery- approximately 15-20 minutes after induction in the operating room (OR)
  blood will be drawn from peripheral venous line, arterial line, and/or central venous line then pH blood value will be assessed by using a bedside point-of-care device, called i-stat.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Tobias, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided